CLINICAL TRIAL: NCT05276063
Title: A Phase 2b, Randomized, Double-Mask, Placebo-Controlled, Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Linsitinib in Subjects With Active, Moderate to Severe Thyroid Eye Disease (TED)
Brief Title: A Phase 2b, Study of Linsitinib in Subjects With Active, Moderate to Severe Thyroid Eye Disease (TED)
Acronym: LIDS
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sling Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGN-TED-301
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Eye Disease; Graves Orbitopathy; Endocrine System Diseases; Eye Diseases; Thyroid Associated Ophthalmopathy; Graves Ophthalmopathy; Thyroid Diseases; Orbital Diseases; Proptosis; IGF1R; Exophthalmos; Hashimoto
Keywords: Thyroid Associated Ophthalmopathies
MeSH Terms: conditions — Graves Ophthalmopathy; Endocrine System Diseases; Eye Diseases; Thyroid Diseases; Orbital Diseases; Exophthalmos; Hashimoto Disease | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo Arm
  Interventions: Drug: Placebo
- Low Dose (Active Comparator): Active Arm Low Dose Linsitinib
  Interventions: Drug: Linsitinib
- High Dose (Active Comparator): Active Arm High Dose Linsitinib
  Interventions: Drug: Linsitinib

INTERVENTIONS:
Drug: Linsitinib — Study medication taken twice daily by mouth
  Arms: High Dose; Low Dose
Drug: Placebo — Placebo taken twice daily by mouth
  Arms: Placebo

SUMMARY:
The overall objective is to study the safety, pharmacokinetics and efficacy of linsitinib (a small molecule IGF-1R inhibitor) administered orally twice daily (BID) vs. placebo, at 24 weeks in the treatment of subjects with active, moderate to severe thyroid eye disease (TED).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Graves' Disease and/or autoimmune Hashimoto's thyroiditis associated with active moderate to severe TED with a CAS ≥ 4 (on the 7- item scale) for the most severely affected eye (primary study eye) at Screening and Baseline
* Confirmed active TED (not sight-threatening but has an appreciable impact on daily life, with onset (as determined by patient records) within 12 months prior to the Baseline visit and usually associated with one or more of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal for race and gender, and/or inconstant or constant diplopia.
* Subjects must be euthyroid with the participant's baseline disease under control or have mild hypo- or hyperthyroidism (defined as free thyroxine [FT4] and free triiodothyronine levels [FT3] < 50% above or below the normal limits) at Screening.
* Does not require immediate ophthalmic surgery, radiotherapy to orbits or other ophthalmological intervention at the time of Screening and is not planning for any such treatment during the course of the study.

Exclusion Criteria:

* Decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months.
* Corneal decompensation unresponsive to medical management.
* Previous orbital irradiation or orbital surgery.
* Any glucocorticoid use (intravenous [IV] or oral) with a cumulative dose equivalent to >= 1g of methylprednisolone or equivalent for the treatment of TED within 3 months of Screening.
* Prior IGF-1R inhibitor therapy for any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Subjects who are Proptosis Responders at Week 24 | 24 weeks

SECONDARY OUTCOMES:
Change from Baseline in Proptosis to Week 24 (Study Eye) | 24 weeks
Percentage of Subjects who are Diplopia Responders at Week 24 | 24 weeks
Percentage of Subjects who are Overall Responders at Week 24 | 24 weeks
Percentage of Subjects who are CAS Categorical Responders at Week 24 (Study Eye) | 24 weeks
Change from Baseline in the Graves' Ophthalmopathy Quality of Life (GO-QoL) Questionnaire Overall Score to Week 24. | 24 weeks

CONTACTS AND LOCATIONS:
Locations (30):
- United States (19):
  - Thrive Health Research, Beverly Hills, California
  - UC San Diego Health, La Jolla, California
  - UCLA, Los Angeles, California
  - Byers Eye Institute - Stanford University, Palo Alto, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Center for Excellence in Eye Care, Miami, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Chicago Oculofacial Plastic Surgery, Chicago, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Mass Eye and Ear, Boston, Massachusetts
  - Kellogg Eye Center, Ann Arbor, Michigan
  - Kahana Oculoplastic & Orbital Surgery, Livonia, Michigan
  - Washington University in St. Louis/Barnes Jewish Hospital, Creve Coeur, Missouri
  - Columbia University, New York, New York
  - Wake Forest Baptist Health Eye Center, Winston-Salem, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Neuro-Eye Clinical Trials, Inc., Bellaire, Texas
  - Eyelid Center of Utah, Salt Lake City, Utah
  - West Virginia University Eye Institute, Morgantown, West Virginia
- Canada (2):
  - Vancouver Coastal Health Eye Care Center, Vancouver, British Columbia
  - Toronto Retina Institute, North York
- Italy (3):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Endocrinology Pawilione Zonda, Milan
  - AOU Pisana, Pisa
  - University of Pisa, Pisa
- Spain (3):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
- United Kingdom (3):
  - Frimley Health Foundation Trust, Camberley
  - Cardiff University, Cardiff
  - Moorfields Eye Hospital NIHR Clinical Research Facility, London

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data collected during the trial, after deidentification will be made available.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to info@slingtx.com